CLINICAL TRIAL: NCT07369440
Title: Community-based Power Training in Faller and Non-faller Older Adults: a Feasibility and Fall Risk Study.
Acronym: POWER-AEQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other)
Responsible Party: Principal Investigator, Óscar Júnio da Silva Ribeiro Requestor Affiliation: Doctor, Doctoral Student, University of Maia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: Ethics committee: 160/2023; 2023.04264.BD (Other Grant/Funding Number: Foundation for Science and Technology (FCT))
Record Dates: First submitted 2024-09-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Fall Prevention; Muscle Power Performance; Functional Mobility; Balance Control in Elderly
Keywords: Older adults; Fallers; Power Training; Functional mobility; Balance

STUDY DESIGN:
Intervention Model Description: The present project will have a randomized study design with delayed onset with an equal number of elderly individuals with and without a history of falls distributed across the intervention groups.
  Participants will be tested initially (PRE_Control), after 12 weeks of control period (PRE_Intervention), after 12 weeks of intervention (POST_Intervention), and after 6 months of follow-up (RET).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional Resistance Training in Older Fallers (Experimental): Retrospective falls incidence of the 12 months prior to enrollment will be used to divide participants into non_fallers (n=60) and fallers (n=60) In this arm of the study, 30 older fallers will perform a multicomponent exercise program focusing on traditional resistance training.
  Interventions: Behavioral: Multi-component exercise program focused on traditional resistance training
- Traditional Resistance Training in Older Non-Fallers (Experimental): Retrospective falls incidence of the 12 months prior to enrollment will be used to divide participants into non_fallers (n=60) and fallers (n=60) In this arm of the study, 30 older non-fallers will perform a multicomponent exercise program focusing on traditional resistance training.
  Interventions: Behavioral: Multi-component exercise program focused on traditional resistance training
- Power Training in Older Fallers (Experimental): Retrospective falls incidence of the 12 months prior to enrollment will be used to divide participants into non_fallers (n=60) and fallers (n=60) In this arm of the study, 30 older fallers will perform a multicomponent exercise program focusing on power training.
  Interventions: Behavioral: Multi-component exercise program focused on muscle power
- Power Training in Older Non-Fallers (Experimental): Retrospective falls incidence of the 12 months prior to enrollment will be used to divide participants into non_fallers (n=60) and fallers (n=60) In this arm of the study, 30 older non-fallers will perform a multicomponent exercise program focusing on power training.
  Interventions: Behavioral: Multi-component exercise program focused on muscle power

INTERVENTIONS:
Behavioral: Multi-component exercise program focused on muscle power — The intervention will be applied for 12 weeks, with a frequency of 3 times per week. Each session will have 45 minutes, and the participants will be instructed to perform a warm-up on a treadmill or other cardiofitness equipment, power training, and balance exercise.
  Participants in the power training groups (30 non-fallers and 30 fallers) will perform knee extension, hip extension and hip abduction exercises, in a regimen of 3 sets of 10 repetitions at 50% of the participant's 1 repetition maximum (1RM), performing each repetition as fast as possible on variable resistance machines. The 1RM estimation will be determined using a 10RM protocol and applying Brzycki's equation. The 1RM assessment will be conducted during the first training session and will be reassessed every 3 weeks to progressively adjust resistance training loads.
  The progression on the balance exercise (stepping and manipulation of the centre of mass over the base of support) will be equally performed every 3 weeks.
  Other Names: Power Training
  Arms: Power Training in Older Fallers; Power Training in Older Non-Fallers
Behavioral: Multi-component exercise program focused on traditional resistance training — The intervention will be applied for 12 weeks, 3 times per week. Each session will have 45 minutes, and the participants will be instructed to perform a warm-up on a cardiofitness equipment, resistance exercise, and balance exercise.
  Participants in the traditional resistance training groups (30 non-fallers and 30 fallers) will perform knee extension, hip extension and hip abduction exercises, in a regimen of 3 sets of 10 repetitions at 60-75% of the participant's 1 repetition maximum (1RM), at a cadence of 2s concentric and 2s eccentric on variable resistance machines. The 1RM estimation will be determined using a 10RM protocol and applying Brzycki's equation. The 1RM assessment will be conducted during the first training session and will be reassessed every 3 weeks to progressively adjust resistance training loads.
  The progression on the balance exercise (stepping and manipulation of the centre of mass over the base of support) will be equally performed every 3 weeks.
  Other Names: Traditional Resistance Exercise
  Arms: Traditional Resistance Training in Older Fallers; Traditional Resistance Training in Older Non-Fallers

SUMMARY:
Aging leads to substantial alterations in the nervous and skeletal muscle systems that ultimately lead to a reduction in "neural drive" and motor performance. While maximal strength starts declining as early as 50 years of age, aging brings even greater reductions in rate of force development and muscle power, that has been shown to be a stronger predictor of functional independence and balance impairments.

Falls are a major health concern as one third of adults over 65 years loses balance and falls every year, and based on a published report, the estimated health care costs associated with falls in the European Union is €25 billion.

The ability to recover balance declines with aging, where older individuals often recover balance with a greater number of balance recovery steps and non-optimal stepping strategies. In addition, older adults have more difficulty recovering balance in the medio-lateral direction. The hip abductors are fundamental in controlling the motion of the body centre of mass in this direction during weight transfers of standing, stepping, and walking.

Furthermore, these muscles appear to be more susceptible to age-related composition and performance declines than other muscles of the lower limbs, especially in individuals at a higher risk for falls.

Unfortunately, common balance interventions, such as, functional balance training, Tai-Chi, or dance, have a very limited capacity to reduce the risk of falls in older adults. Interestingly, resistance training is relatively better than the mentioned interventions at reducing this problem. This may come about through mitigating the agerelated neuromuscular performance deficits. However, traditional resistance training lacks the emphasis in high velocity movements required for adequate fall prevention protective stepping strategies. Muscle power training is a safe and effective alternative to traditional resistance training. By emphasizing in maximum speed of execution, its results are often better than with traditional resistance training, especially in functional outcomes, with the potential to enhance balance recovery. However, there is little and inconsistent evidence on the optimal exercise parameters (such as velocity) for prevention of falls.

Community-based multi-component exercise programs are often used to promote health and functional benefits in the older adult population. These programs not only have a positive impact in a larger number of communitydwelling individuals, but can also lead to significant improvements. Nonetheless, these programs limited in reducing the risk for falls. Considering the robust effects of muscle power training in the older population, it is conceivable that a multi-component community-based exercise intervention, that focuses on developing muscle power and reduce fall risk, can improve the older individuals' ability to recover balance and consequently, bring greater benefits to the older adult community. However, there is no information on the feasibility of conducting an exercise program to develop muscle power and reduce fall risk in a community-based setting. Furthermore, it is generally unknown if such an exercise intervention can improve function, balance, and reduce the occurrence of falls in older adults especially, among those that have fallen in the past- which are the most relevant target population for both clinical studies and practice.

DETAILED DESCRIPTION:
This study will adopt a randomized controlled trial design comparing a community-based multi-component exercise program focused on muscle power (MCP) with a traditional community-based multi-component exercise program (TMC). Equal numbers of older adults with and without a history of falls will be allocated to each intervention group.

1. Participants

   Based on the effect size calculated (0.55-1.75), to achieve a statistical power of 80% with a significance of p smaller than 0.05, this study would need to recruit approximately 22 subjects per group. Anticipating 20% dropout and attrition, and considering this study will propose four different groups, a total of 120 community-dwelling older adults will be recruited from the greater Porto area through existing partnerships with Maia's municipality. Retrospective falls incidence during the 12 months prior to enrollment will be used to classify participants as fallers (n=60) or non-fallers (n=60). Using stratified randomization, participants will be allocated to one of four groups: TMC non-fallers (n=30), TMC fallers (n=30), MCP non-fallers (n=30), or MCP fallers (n=30).

   The study will be conducted in accordance with the Declaration of Helsinki of 1975, revised in 2013 and General Data Protection Regulation (GDPR) requirements. Ethical approval will be obtained from the Ethics Committee of the University of Maia prior to participant enrollment. Written informed consent will be obtained from all participants before participation.
2. Procedures

   2.1.Screening

   An initial screening will ascertain if participants meet the inclusion/exclusion criteria. Additionally, the International Physical Activity Questionnaire will be applied to control for physical activity as confounding factor.

   2.2.Assessments

   Pre_Control, Pre_Intervention, Post_Intervention and Ret sessions will be identical and will consist of functional mobility and balance tests, including gait speed, mini-BESTest, Four Square Step Test (FSST) and five time Sit-to-Stand (5STS) test. Neuromuscular assessments, consisting of isometric maximal voluntary contractions (IMVC) of the handgrip (Gripwisetech, PT), knee extensors, hip extensors and hip abductors (DESMOTEC, IT), at a collection frequency of 100Hz. Participants will be instructed to "push as hard and as fast as possible" for 15 seconds.

   A questionnaire assessing participant perspectives on the exercise intervention will be used at week 13. Adverse events and falls incidence will be assessed monthly via questionnaire from Pre_Control-Ret.
3. Interventions

   TMC and MCP interventions will be applied for 12 weeks, 3 times per week. Both interventions will be composed by aerobic exercises, such as walking overground and/or on a treadmill at the preferred speed, balance exercises involving stepping and manipulation of the center of mass over the base of support and resistance training. In the resistance training, participants will perform knee extension, hip extension and hip abduction exercises, in a regimen of 3 sets of 10 repetitions at 60-75% of the participant's 1 repetition maximum (1RM), with weights and/or weight machines. 1RM estimation will be done through a 10RM protocol and apply Brzycki's equation. 1RM assessment will be conducted on the first training session and re-done every 3 weeks to progressively adjust resistance training loads.

   While in TMC participants will be instructed to perform the repetitions of the resistance exercises at a cadence of 2s concentric and 2s eccentric, participants in the MCP will be instructed to perform every repetition as fast as possible. To maintain high velocity in this group, 50% of 1RM training load will used.
4. Statistical Analyses

   A linear mixed effects model will test the main effects of intervention, group and time, and their interactions, for a significance level of p less than 0.05.
5. Expected outcomes

   The interventions are expected to be feasible and safe and it will have a positive adherence.Therefore, the application of muscle power training within a community-based multi-component setting is expected to be feasible.

   The muscle power-focused multi-component exercise program (MCP) is expected to produce greater improvements in neuromuscular performance and functional mobility when compared to the traditional multi-component exercise program (TMC).

   Participants with a history of falls are expected to demonstrate larger relative improvements in neuromuscular and functional outcomes compared to non-fallers, due to greater baseline impairments.

   Improvements achieved following the MCP intervention are expected to be maintained over time and associated with a reduction in falls incidence during the post-intervention follow-up period.
6. Potential risks and contingency plans

Multi-component exercise programs, including muscle power-oriented training, have been previously applied safely in community-dwelling older adults. Therefore, the risk of adverse effects associated with the TMC and MCP interventions is considered low.

Participant safety will be monitored throughout the study, and any adverse symptoms or events will be documented and addressed accordingly.

There is a possibility that the interventions may not result in statistically significant improvements. In the event that observed effect sizes are smaller than anticipated, the lack of significant differences may be attributable to sample size limitations. In such cases, recruitment may be extended to increase the study sample.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65-85 years;
* Fall history over the 12 months prior to enrollment (fallers group).

Exclusion Criteria:

* Any existing medical conditions or injuries which would affect the ability or safety to perform exercise;
* Taking medication affecting balance (such as sedatives, anti-depressives);
* Regular (more than 1d/week) participation in resistance training with loading greater than bodyweight during the last year;
* BMI greater than 32 kg/m2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular Assessments | 12 weeks
  Handgrip strength was assessed through sustained isometric maximal voluntary contractions (IMVC) using a digital handgrip dynamometer (Gripwisetech, PT). Participants were seated with the shoulder adducted, elbow flexed at 90°, forearm in neutral position and wrist in slight extension. Three maximal isometric contractions of 15 seconds were performed with the dominant hand, with 2 minutes of rest between trials. Maximal force was defined as the highest peak force achieved during the contraction. Rate of force development (RFD) was calculated as the slope of the force-time curve during the initial phase of contraction (0-200 ms). The best trial was used for analysis.
Neuromuscular Assessments | 12 weeks
  Maximal isometric strength of the knee extensors, hip extensors, and hip abductors was assessed using isometric maximal voluntary contractions (IMVC) with a computer-controlled dynamometer (DESMOTEC, IT). All contractions were performed at the joint neutral position (0°) defined for each test. Participants performed the tests in a seated position for knee extension and in a standing position for hip extension and hip abduction, using standardized testing positions. For each muscle group, three maximal isometric contractions of 15 seconds were performed, with 2 minutes of rest between trials. Maximal force was defined as the highest peak torque achieved during the contraction. Rate of force development (RFD) was calculated from the slope of the torque-time curve during the initial phase of the contraction (0-200 ms). The best trial was used for analysis. Data were sampled at 100 Hz.
Functional Mobility and Balance | 12 weeks
  Time to complete four meters at the preferred gait speed (4MWT).
Functional Mobility and Balance | 12 weeks
  Time to complete the Four Square Step Test (FSST).
Functional Mobility and Balance | 12 weeks
  Time to stand up and sit down five times (5STS) as quickly as possible.
Functional Mobility and Balance | 12 weeks
  Total score of the Mini-BESTest (0-28 points).
Functional Mobility (TUG). | 12 weeks
  Time to complete the Timed Up and Go test (seconds).
Functional Mobility under Dual Task | 12 weeks
  Time to complete the Timed Up and Go test under dual-task conditions (seconds).

SECONDARY OUTCOMES:
Feasibility (Recruitment Rate) | 12 weeks
  Proportion of eligible participants who were enrolled in the study, expressed as a percentage (%).
  The analysis of feasibility and safety of the interventions will include recruitment rate, adherence to the intervention, and adverse events.
Feasibility (Intervention Adherence) | 12 weeks
  Percentage of prescribed intervention sessions attended by participants during the intervention period (%).
  The analysis of feasibility and safety of the interventions will include recruitment rate, adherence to the intervention, and adverse events.
Safety (Adverse Events) | 12 weeks
  Number and type of adverse events collected monthly through a structured questionnaire during both the control period and the intervention period.
  The analysis of feasibility and safety of the interventions will include recruitment rate, adherence to the intervention, and adverse events.
Prospective falls incidence | 6 months
  Prospective falls incidence will be recorded as the number of unintentional falls occurring during the 6 months between Post-Ret.

CONTACTS AND LOCATIONS:
Locations (1):
- Maia Municipal Sports Hall, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Kotob R, Giangregorio LM. Pilot and feasibility studies in exercise, physical activity, or rehabilitation research. Pilot Feasibility Stud. 2018 Aug 14;4:137. doi: 10.1186/s40814-018-0326-0. eCollection 2018. PMID 30123527
- [Background] Munoz-Bermejo L, Adsuar JC, Mendoza-Munoz M, Barrios-Fernandez S, Garcia-Gordillo MA, Perez-Gomez J, Carlos-Vivas J. Test-Retest Reliability of Five Times Sit to Stand Test (FTSST) in Adults: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Jun 9;10(6):510. doi: 10.3390/biology10060510. PMID 34207604
- [Background] Lane C, McCrabb S, Nathan N, Naylor PJ, Bauman A, Milat A, Lum M, Sutherland R, Byaruhanga J, Wolfenden L. How effective are physical activity interventions when they are scaled-up: a systematic review. Int J Behav Nutr Phys Act. 2021 Jan 22;18(1):16. doi: 10.1186/s12966-021-01080-4. PMID 33482837
- [Background] Sherrington C, Whitney JC, Lord SR, Herbert RD, Cumming RG, Close JC. Effective exercise for the prevention of falls: a systematic review and meta-analysis. J Am Geriatr Soc. 2008 Dec;56(12):2234-43. doi: 10.1111/j.1532-5415.2008.02014.x. PMID 19093923
- [Background] Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JCT, Lord SR. Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(24):1750-1758. doi: 10.1136/bjsports-2016-096547. Epub 2016 Oct 4. PMID 27707740
- [Background] Robinovitch SN, Feldman F, Yang Y, Schonnop R, Leung PM, Sarraf T, Sims-Gould J, Loughin M. Video capture of the circumstances of falls in elderly people residing in long-term care: an observational study. Lancet. 2013 Jan 5;381(9860):47-54. doi: 10.1016/S0140-6736(12)61263-X. Epub 2012 Oct 17. PMID 23083889
- [Background] Mille ML, Johnson-Hilliard M, Martinez KM, Zhang Y, Edwards BJ, Rogers MW. One step, two steps, three steps more ... Directional vulnerability to falls in community-dwelling older people. J Gerontol A Biol Sci Med Sci. 2013 Dec;68(12):1540-8. doi: 10.1093/gerona/glt062. Epub 2013 May 17. PMID 23685768
- [Background] Hartholt KA, Polinder S, Van der Cammen TJ, Panneman MJ, Van der Velde N, Van Lieshout EM, Patka P, Van Beeck EF. Costs of falls in an ageing population: a nationwide study from the Netherlands (2007-2009). Injury. 2012 Jul;43(7):1199-203. doi: 10.1016/j.injury.2012.03.033. Epub 2012 Apr 27. PMID 22541759
- [Background] Metter EJ, Conwit R, Tobin J, Fozard JL. Age-associated loss of power and strength in the upper extremities in women and men. J Gerontol A Biol Sci Med Sci. 1997 Sep;52(5):B267-76. doi: 10.1093/gerona/52a.5.b267. PMID 9310077
- [Background] Fielding RA, LeBrasseur NK, Cuoco A, Bean J, Mizer K, Fiatarone Singh MA. High-velocity resistance training increases skeletal muscle peak power in older women. J Am Geriatr Soc. 2002 Apr;50(4):655-62. doi: 10.1046/j.1532-5415.2002.50159.x. PMID 11982665
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Mehmet H, Robinson SR, Yang AWH. Assessment of Gait Speed in Older Adults. J Geriatr Phys Ther. 2020 Jan/Mar;43(1):42-52. doi: 10.1519/JPT.0000000000000224. PMID 30720555
- [Background] Inacio M, Creath R, Rogers MW. Low-dose hip abductor-adductor power training improves neuromechanical weight-transfer control during lateral balance recovery in older adults. Clin Biomech (Bristol). 2018 Dec;60:127-133. doi: 10.1016/j.clinbiomech.2018.10.018. Epub 2018 Oct 13. PMID 30343209
- [Background] Reid KF, Callahan DM, Carabello RJ, Phillips EM, Frontera WR, Fielding RA. Lower extremity power training in elderly subjects with mobility limitations: a randomized controlled trial. Aging Clin Exp Res. 2008 Aug;20(4):337-43. doi: 10.1007/BF03324865. PMID 18852547
- [Background] Lopes PB, Pereira G, Lodovico A, Bento PC, Rodacki AL. Strength and Power Training Effects on Lower Limb Force, Functional Capacity, and Static and Dynamic Balance in Older Female Adults. Rejuvenation Res. 2016 Oct;19(5):385-393. doi: 10.1089/rej.2015.1764. Epub 2016 Mar 3. PMID 26707497
- [Background] Inacio M, Ryan AS, Bair WN, Prettyman M, Beamer BA, Rogers MW. Gluteal muscle composition differentiates fallers from non-fallers in community dwelling older adults. BMC Geriatr. 2014 Mar 25;14:37. doi: 10.1186/1471-2318-14-37. PMID 24666603
- [Background] Rogers MW, Mille ML. Lateral stability and falls in older people. Exerc Sport Sci Rev. 2003 Oct;31(4):182-7. doi: 10.1097/00003677-200310000-00005. PMID 14571957
- [Background] Kallman DA, Plato CC, Tobin JD. The role of muscle loss in the age-related decline of grip strength: cross-sectional and longitudinal perspectives. J Gerontol. 1990 May;45(3):M82-8. doi: 10.1093/geronj/45.3.m82. PMID 2335723
- [Background] Aagaard P, Suetta C, Caserotti P, Magnusson SP, Kjaer M. Role of the nervous system in sarcopenia and muscle atrophy with aging: strength training as a countermeasure. Scand J Med Sci Sports. 2010 Feb;20(1):49-64. doi: 10.1111/j.1600-0838.2009.01084.x. PMID 20487503
- See also: Strength Testing-Predicting a One-Rep Max from Reps-to-Fatigue — https://www.researchgate.net/publication/273371811_Strength_Testing-Predicting_a_One-Rep_Max_from_Reps-to-Fatigue
- See also: The Loss of Power and Need for Power Training in Older Adults — https://www.academia.edu/94778131/The_Loss_of_Power_and_Need_for_Power_Training_in_Older_Adults?uc-sb-sw=34431134